CLINICAL TRIAL: NCT04817956
Title: Improving Public Cancer Care by Implementing Precision Medicine in Norway A Multi-cohort Phase 2 Treatment Clinical Study Investigating Efficacy of Approved Drugs Outside Indication in Patients With Advanced Cancer
Brief Title: Improving Public Cancer Care by Implementing Precision Medicine in Norway
Acronym: IMPRESS-N
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); Hospital of Southern Norway Trust (Other); Ostfold Hospital Trust (Other); The Hospital of Vestfold (Other); Helse Stavanger HF (Other Government); Nordlandssykehuset HF (Other); Sykehuset Innlandet HF (Other); Helse Forde (Other); Helse Fonna (Other); Helse Nord-Trøndelag HF (Other); Helse Møre og Romsdal HF (Other Government); Sykehuset Telemark (Other Government); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Åslaug Helland, Research Leader, Oncologist, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPRESS-Norway
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cancer Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — atezolizumab; Bevacizumab; alectinib; HhAntag691; entrectinib; Vemurafenib; niraparib; dostarlimab; ceritinib

STUDY DESIGN:
Intervention Model Description: Simon 2-stage Basket-Umbrella
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (20):
- Atezolizumab (Experimental): Atezolizumab used outside of current indication, based on biomarkers
  Interventions: Drug: Atezolizumab
- Atezilizumab combined with bevacizumab (Experimental): Atezilizumab combined with bevacizumab used outside of indication, based on biomarkers
  Interventions: Drug: Atezolizumab
- Phesgo (trastuzumab og pertuzumab) (Experimental): Phesgo used outside of indication, based on biomarkers.
  Interventions: Drug: Atezolizumab
- Alectinib (Experimental): Alectinib used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- vismodegib (Experimental): vismodegib used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- entrectinib (Experimental): entrectinib used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- Zelboraf + Cotellic (Experimental): Zelboraf + Cotellic used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- Alpelisib (Experimental): Alpelisib used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- Dabrafenib + trametinib (Experimental): Used outside of indication, based on biomarker
  Interventions: Drug: Atezolizumab
- Melfalan (Experimental): Melfalan used outside ofcurrent indication
  Interventions: Drug: Atezolizumab
- Pemazyre (Experimental): Pemazyre used outside ofcurrent indication
  Interventions: Drug: Atezolizumab
- Selpercatinib (Experimental): used outside ofcurrent indication
  Interventions: Drug: Atezolizumab
- Olaparib (Experimental): Used outside of current indication, for patients with bi-allelic BRCA-inactication
  Interventions: Drug: Atezolizumab
- Capmatinib (Experimental): Used outside of current indication,
  Interventions: Drug: Atezolizumab
- Imatinib (Experimental): Used outside of current indication,
  Interventions: Drug: Atezolizumab
- Bortezomib (Experimental): Used outside of current indication,
  Interventions: Drug: Atezolizumab
- Actinomycin D (Experimental): Used outside of current indication,
  Interventions: Drug: Atezolizumab
- Niraparib (Experimental): Used outside of current indication,
  Interventions: Drug: Atezolizumab
- Dostarlimab (Experimental): Used outside of current indication
  Interventions: Drug: Atezolizumab
- Ceritinib (Experimental): Used outside of current indication
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — drugs used outside indication, based on biomarker
  Other Names: Atezolizumab combined with bevacizumab; Phesgo (trastuzumab og pertuzumab); Alectinib; vismodegib; entrectinib; Vemurafenib and cobemitinib; Niraparib; Dostarlimab; Ceritinib

SUMMARY:
IMPRESS-Norway is a prospective, non-randomized clinical trial evaluating efficacy of commercially available, anti-cancer drugs prescribed for patients with advanced cancer diagnosed with potentially actionable alterations as revealed by molecular diagnostics. IMPRESS-Norway is a nation-wide study and all hospitals with an oncology and / or hematology department will be invited to participate in the study. The study will use a combined umbrella and basket design and a Simon two-stage model of expanding cohorts to follow up potentially effective combinations of biomarker and drug on specific indications. Sampling of biological material will be performed at presentation, during treatment and upon progression. Additional biomarker and translational analyses including whole genome sequencing (WGS) on tumour material and liquid biopsies, identifying mechanisms underlying drug sensitivity versus resistance will be performed.

DETAILED DESCRIPTION:
Eligible patients have an advanced malignancy already treated with standard treatment, acceptable performance status and organ function, with no other suitable clinical trial available in Norway. A molecular test performed at a study specific reference laboratory has identified a potentially targetable molecular profile. Next, a suitable drug should be available from the trial drug armamentarium. Finally, if the patient fulfils the inclusion criteria and is accepted for the trial, a second tumour biopsy (snap-frozen)/ tumour material for WGS will be sampled. Patients enrolled in the study will enter an existing cohort, or, in case a suitable cohort does not exist, a new cohort can be opened. One cohort will consist of one diagnostic subgroup, one drug (or one drug-combination) and one molecular marker. The choice of drug(s) will be supported by a list of potential profiles. In addition, available knowledge from the literature will be used to prepare discussion in a national molecular tumour board, which will provide a treatment recommendation to the treating physician and the study doctors . The protocol-specified treatment may be administered to the patient once drug-specific eligibility criteria are confirmed and a fresh pre-treatment biopsy is performed for future biomarker studies and research on responders versus non-responders.

All patients who receive treatment with a drug available in the protocol will be monitored for standard efficacy outcomes including tumour response, progression-free and overall survival as well as study specific measures as duration of treatment. Patients that are screened, but not included into any cohorts will be followed for 16 weeks for survival and clinical course of disease. Treatment-related toxicities (CTCAE grade 3-5) will be evaluated. Study-specific treatment and outcome data including results from the molecular screening will be reported to the Cancer Registry of Norway. Long-term follow up data using the Cancer Registry of Norway and information from The Norwegian Patient Registry, The Norwegian Prescription Database and Primary patient- and user Register (KPR) will be collected on all patients screened.

ELIGIBILITY:
Inclusion Criteria:

* Type of Participant and Health status

  1. Patient with a pathology-proven locally advanced or metastatic malignant disease who is no longer benefitting from standard anti-cancer treatment or for whom, in the opinion of the investigator, no such treatment is available or indicated.
  2. ECOG performance status 0-2.
  3. For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
  4. Patients must have acceptable organ function as defined below. However, as noted above, drug-specific inclusion/exclusion criteria specified in the drug-specific study manuals for each agent will take precedence for this and all inclusion criteria (exceptions for haematological diagnoses):

     1. Absolute neutrophil count ≥ 1.5 x109 / L
     2. Hemoglobin > 9 g/dl
     3. Platelets > 75,000/µl
     4. Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
     5. AST (SGOT) and ALT(SGPT) < 2.5 x institutional upper limit of normal (ULN) (or < 5 x ULN in patients with known hepatic metastases)
     6. Calculated or measured creatinine clearance ≥ 40 mL/min/1.73 m2.
  5. Patients must have measurable or evaluable disease. RECIST v1.1 (10, 18) will be used for patients with solid tumours. For patients with multiple myeloma or non-Hodgkin lymphoma, IMWG response criteria (19) and CHESON/Lugano guidelines (20) will be used, resp. For glioblastoma patients, RANO criteria will be used (21). iRECIST will be used for immunotherapy-cohorts. IWG response criteria will be used for haematological cancers.

     Patients whose disease cannot be objectively measured by physical or radiographic examination (e.g., elevated serum tumour marker only) are NOT eligible, with the exception of CA-125 for ovarian cancer and PSA for prostate cancer (22).
  6. Results must be available from a genomic / molecular test performed in a preapproved laboratory (Section 10.15). The test used to qualify a patient for participation in IMPRESS-Norway may have been performed on any specimen of the patient's tumour obtained at any point during the patient's care at the discretion of the patient's treating physician. Genomic assays performed on cell-free DNA in plasma ("liquid biopsies") will also be acceptable if the genomic analysis is performed as defined in Section 10.5. NGS analyses will be performed on a newly sampled biopsy if possible. Information from these analyses might be used upon progression, for evaluation of possible new cohort-inclusion.
  7. Have a genomic profile for which treatment with one of the approved targeted anti-cancer therapies included in this study has potential clinical benefit see Section 4.3.5

     Note: Eligible genomic tests may include any of the following technologies and equivalent techniques: Immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR) (incl nanostring), array-based copy number analysis (CNV), sanger sequencing (SS), RNA sequencing, gene panels or whole exome sequencing (WES) by next generation sequencing (NGS). The test may have been performed on a fresh (frozen or in RNA-later) or paraffin-embedded specimen of the primary tumour or a metastatic deposit or on cell-free DNA derived from liquid biopsies (like for instance peripheral blood plasma), as determined by the treating physician, and must reveal a potentially actionable genomic variant or protein overexpression as defined in Section 4.3.
  8. Patients must meet drug-specific eligibility requirements for the drug selected by the investigator.

Sex and Contraceptive/Barrier Requirements 9.8. Because of the risks of drug treatment to the developing fetus, women of child-bearing potential and men must agree to use adequate highly effective methods of contraception for the duration of study participation, and for 4 to 24 months following completion of study therapy as defined in Section 11.4.

10.9. Female participants must have a negative highly sensitive pregnancy test <1 month prior to inclusion.

11.10. Male patients should avoid impregnating a female partner. Male study patients must agree to one of the following: practice effective barrier contraception as described under sec. 11.4 during the entire study treatment period and through a certain time after the last dose of study drug. Details are given in the "Drug specific amendment".

Informed Consent 12.11. Ability to understand and the willingness to sign a written informed consent/assent document as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Guardians / parents can act on behalf of children.

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study (other exclusion criteria might apply for specific drugs).

Medical Conditions

1. Patients eligible to enter other ongoing trials which have to potential to benefit the patients equally or more than a IMPRESS-Norway cohort, and for whom access to the ongoing trials is manageable (taking geography into consideration).
2. Ongoing toxicity > CTCAE grade 2, other than peripheral neuropathy, related to anti-tumour treatment that was completed within 4 weeks prior to treatment initiation. Patients with ongoing peripheral neuropathy of ≥ CTCAE grade 3.

   Patients with known progressive brain metastases determined by serial imaging or declining neurologic function in the opinion of the treating physician. Patients with previously treated / stable brain metastases are eligible. Additional exclusion criteria specific for GBM patients:

   a. Patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs (non-EIAED). EIAED are prohibited. Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to randomization.
3. Patients with the following pre-existing cardiac conditions, uncontrolled angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure.
4. Patients with left ventricular ejection fraction (LVEF) known to be < 40%.
5. Patients with stroke (including TIA) or acute myocardial infarction within 4 months before the first dose of study treatment
6. Patients with acute gastrointestinal bleeding within 1 month of start of treatment
7. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, severe psychiatric illness situations, or anticipated or planned anti-cancer treatment or surgery.
8. Patients with known allergy/hypersensitivity to the study drug (active substance or to any of the excipients).

Prior/Concomitant Therapy 9. Previous treatment with the selected study drug for the same malignancy. 10. Patient is receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g., megestrol acetate, bisphosphonates) or ongoing castration-intent therapy for prostate cancer. These medications must have been started ≥ 1 month prior to enrolment on this study. Patients may be on warfarin, low molecular weight heparin or direct factor Xa inhibitors, unless such therapies are prohibited by drug-specific exclusion criteria.

Diagnostic assessments 11. If the patient's tumour has a genomic variant known to confer resistance to an anti-cancer agent available in this study, the patient will not be eligible to receive that agent but will be eligible to receive other drugs available in this study if all inclusion and exclusion criteria are met for that drug.

Other Exclusions 12. Female patients who are pregnant or nursing 13. Patients who do not meet drug-specific eligibility requirements for the drug selected by the investigator

Note: For each drug included in this protocol, specific inclusion and exclusion criteria (based on the Summary of Product Characterics (SPC) or manufacturer's recommendations) may also apply. These can be found in the supplemental information about each agent included in the appendices. Drug-specific inclusion and exclusion criteria will take precedence over the general inclusion/exclusion criteria

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2040-03-30 (Estimated); Study Completion 2045-04-30 (Estimated)

PRIMARY OUTCOMES:
16 weeks clinical response | 16 weeks
  To determine percentage of patients who have "not progression" on treatment. "Not progression" is complete response, partial response and stable disease.
Access to drugs for patients | 4 years
  To evaluate percentage of patients included in treatment cohorts

SECONDARY OUTCOMES:
Progression free survival of patients starting treatment in the study | 4 years
  Progression-free survival
  Time from treatment initiation to progression of disease
Overall survival of patients starting treatment in the study | 4 years
  Time from treatment initiation to death Duration of time on drug Time from the molecular diagnostics first informed consent to starting treatment
Biomarker analyses | 4 years
  • Estimate the percentage of patients eligible for analyses only by liquid biopsies
• Access of tumour tissue biopsy across and within tumour types | 4 years
  • Number of tumour / molecular assessments per patient / cohort

CONTACTS AND LOCATIONS:
Overall Officials: Åslaug Helland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (17):
- Norway (17):
  - Sykehuset Ålesund, Ålesund
  - Haukeland universitetssykehus, Bergen
  - Nordlandssykehuset, Bodø
  - Vestre Viken Hospital, Drammen
  - Førde Hospital, Førde
  - Sykehuset Innlandet, Hamar
  - Helse Fonna, Haugesund
  - Sørlandet sykehus, Kristiansand
  - Sykehuset Levanger, Levanger
  - Oslo University Hospital, Oslo
  - Ahus, Oslo
  - Sykehuset Telemark, Skien
  - Stavanger universitetssykehus, Stavanger
  - Universitetssykehuset i Nord-Norge, Tromsø
  - St Olavs Hospital, Trondheim
  - Sykehuset Vestfold, Tønsberg
  - Sykehuset Østfold Kalnes, Fredrikstad, Østfold fylke

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish results from the study, reporting on our predefined endoints
Supporting Information: CSR
Time Frame: 4 years
Access Criteria: academic interest

REFERENCES:
- [Derived] Helland A, Russnes HG, Fagereng GL, Al-Shibli K, Andersson Y, Berg T, Bjorge L, Blix E, Bjerkehagen B, Brabrand S, Cameron MG, Dalhaug A, Dietzel D, Donnem T, Enerly E, Flobak A, Fluge S, Gilje B, Gjertsen BT, Gronberg BH, Gronas K, Guren T, Hamre H, Haug A, Heinrich D, Hjortland GO, Hovig E, Hovland R, Iversen AC, Janssen E, Kyte JA, von der Lippe Gythfeldt H, Lothe R, Lund JA, Meza-Zepeda L, Munthe-Kaas MC, Nguyen OTD, Niehusmann P, Nilsen H, Puco K, Ree AH, Riste TB, Semb K, Steinskog ESS, Stensvold A, Suhrke P, Tennoe O, Tjonnfjord GE, Vassbotn LJ, Aas E, Aasebo K, Tasken K, Smeland S. Improving public cancer care by implementing precision medicine in Norway: IMPRESS-Norway. J Transl Med. 2022 May 14;20(1):225. doi: 10.1186/s12967-022-03432-5. PMID 35568909